CLINICAL TRIAL: NCT02059135
Title: Prospective Randomized Double-Blind, Placebo Controlled Evaluation of the Pharmacokinetics, Safety and Efficacy of Recombinant Antithrombin Versus Placebo in Preterm Preeclampsia (PRESERVE-1)
Brief Title: Pharmacokinetics, Safety and Efficacy Study of Recombinant Antithrombin Versus Placebo in Preterm Preeclampsia
Acronym: PRESERVE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: rEVO Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB AT PPE 01-13
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Preterm preeclampsia; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recombinant Human Antithrombin (ATryn) (Active Comparator): ATryn 250 mg loading dose over 15 minutes, immediately followed by continuous infusion of 2000 mg per 24 hours. Total daily dose is 2250 mg for the first day and 2000 mg on subsequent days
  Interventions: Biological: Recombinant human antithrombin (ATryn)
- Normal Saline 0.9% (Placebo Comparator): Placebo (Normal Saline 0.9%, matched for volume of active treatment) consisting of a loading dose over 15 minutes followed by continuous infusion.
  Interventions: Other: Normal Saline 0.9%

INTERVENTIONS:
Biological: Recombinant human antithrombin (ATryn) — Atryn 250 mg loading dose over 15 minutes, immediately followed by continuous infusion of 2000 mg per 24 hours. Total daily dose is 2250 mg for the first day and 2000 mg on subsequent days
  Other Names: Recombinant human antithrombin (rhAT)
  Arms: Recombinant Human Antithrombin (ATryn)
Other: Normal Saline 0.9% — Placebo Comparator: Normal Saline 0.9%
  Other Names: Normal Saline
  Arms: Normal Saline 0.9%

SUMMARY:
The purpose of the study is to assess the efficacy, safety and pharmacokinetics (PK) of recombinant human antithrombin (ATryn) in addition to expectant management for the treatment of preterm preeclampsia (PPE). Efficacy will be assessed by comparing the difference in extension of gestational age from the time of randomization into the study until delivery between ATryn and placebo treated subjects. In addition, the effect of ATryn on fetal and neonatal clinical outcomes will be assessed. The PK characteristics of ATryn in the subjects will be investigated by measuring AT activity levels in the mother during treatment and in cord blood.

DETAILED DESCRIPTION:
Hospitalized PPE patients who are being expectantly managed, after initial assessment and stabilization period, will be considered for the study. After informed consent has been obtained subjects will be screened for eligibility. Screening includes obtaining the subject's medical/obstetric history and a physical examination which includes an assessment of maternal and fetal status. Blood samples for hematology, clinical chemistries, biomarkers, coagulation, immunogenicity and AT activity levels will be drawn. Urine will be collected for baseline urinalysis, protein/creatinine ratio and biomarkers. Eligible subjects who meet inclusion/exclusion criteria will be randomized in a 1:1 ratio to receive a continuous infusion of either ATryn or placebo.

Sampling for AT activity will be performed immediately prior to the first dose of study drug and at specified times thereafter.

Subjects will continue on study drug until maternal and/or fetal indications for delivery necessitate cessation of expectant management or until 34 0/7 weeks of gestation. The average extension of pregnancy with standard of care expectant management in this patient population is approximately 7 days. It is assumed that treatment with ATryn will provide an additional increase in gestational age of 5-7 days as compared to this standard of care. Total duration on study drug is therefore estimated to be approximately 7 to 14 days on average.

Post treatment assessments of the mother will be performed at hospital discharge and approximately 4-6 weeks after delivery of the neonate. Information on the neonates will be collected until they reach a post-menstrual age (PMA) of 36 weeks. If the neonate reaches 36 weeks PMA < 28 days following delivery, the final neonatal follow-up visit should be done at the 4-6 week post-delivery visit.

After the primary study completion and follow-up period, the neonate total number of days in the Neonatal Intensive Care Unit (NICU), days on a ventilator, days requiring supplemental oxygen (FiO2 ≥21%),the neonate hospital discharge date and whether the neonate is discharged from the hospital with a requirement for supplemental home oxygen therapy will be collected to help assess health care utilization. In addition, the date of death will be collected if the neonate expires before hospital discharge. These data will be considered supplemental to the primary study data set.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized female pregnant patients of gestational age of ≥23 0/7 weeks to ≤30 0/7 weeks (for subjects at gestational age 23 0/7 to 23 6/7 all standard interventions including antenatal steroids and cesarean for fetal indications must be offered).

   Gestational age determination by local practice using one of the following three approaches:
   * Last menstrual period (LMP) dating and confirmatory ultrasound
   * Ultrasound alone when LMP is not reliable
   * Known date of conception in the setting of assisted reproductive technology
2. At least 16 years of age (NOTE: different age restrictions may apply per local regulation and/or ethical considerations; subjects under the local age of consent may be excluded at the discretion of the reviewing Institutional Review Board (IRB)
3. Recent diagnosis of Preeclampsia or Superimposed Preeclampsia as defined by:

   • For Preeclampsia
   * Gestational hypertension defined as a recorded systolic blood pressure (BP) of

     ≥140 mm Hg or diastolic BP of ≥90 mm Hg on 2 occasions at least 4 hours apart (since the commencement of medical intervention in any facility) OR
   * Severe gestational hypertension defined as systolic blood pressure of ≥ 160 mm Hg or diastolic blood pressure ≥ 110 mm Hg, confirmed with second assessment within a short interval (minutes) AND
   * New onset of any of the following:

     * Proteinuria defined as ≥0.3 g protein per 24 hours in a 12-24 hour urine collection or protein/creatinine ratio of ≥0.3 mg/mg* (on a random sample or any collection period.)
     * Platelet count less than 100,000/μL
     * Serum creatinine concentrations greater than 1.1 mg/dL in the absence of other renal disease
     * Elevated liver transaminases to ≥ twice upper limit of normal
     * Cerebral or visual symptoms

   For Superimposed preeclampsia:
   * The start of antihypertensive medication, increasing the dose of a currently administered antihypertensive medication or adding a second antihypertensive medication after 20 weeks of pregnancy for systolic BP ≥ 160 or diastolic BP ≥ 105 in a patient that had a previous history of controlled hypertension before 20 weeks of pregnancy. AND
   * New onset of any of the following:

     * proteinuria defined as ≥0.3 g protein per 24 hours in a 12-24 hour urine collection or protein/creatinine ratio of ≥0.3 mg/mg (on a random sample or any collection period)
     * Platelet count less than 100,000/μL
     * Serum creatinine concentrations greater than 1.1 mg/dL in the absence of other renal disease
     * Elevated liver transaminases to ≥ twice upper limit of normal
     * Cerebral or visual symptoms
4. In the opinion of the investigator the patient has demonstrated sufficient clinical stability to be eligible for expectant management
5. The patient is expected to be managed as an inpatient until delivery
6. Signed informed consent for both subject and neonate

Exclusion Criteria:

1. Criteria that would likely require immediate delivery of the fetus are exclusionary if present just prior to randomization:

   * Refractory hypertension despite maximal medical intervention of systolic BP ≥160 mm Hg or diastolic BP of ≥110 mm Hg
   * Thrombocytopenia (platelets ˂ 100/mm3) with or without Hemolysis elevated liver enzymes low platelets (HELLP) syndrome defined as defined as Aspartate amino transferase (AST) ≥70 units/L, and platelets ˂100/mm3, and evidence of hemolysis on blood film plus either Lactic dehydrogenase (LDH) ≥600 IU/mL or total bilirubin ≥1.2 mg/dL)
   * Oliguria (≤500 mL/24 hours) or evidence of progressive renal insufficiency
   * Serum creatinine concentration greater than 1.1 mg/dL
   * Persistent visual disturbances
   * Placental abruption
   * Pulmonary edema
   * Nonreassuring fetal heart rate tracing
   * Intractable headache unrelieved with analgesia
   * Intractable right upper quadrant abdominal pain or vomiting
   * If umbilical Doppler ultrasound has been performed, the presence of an abnormal umbilical artery Doppler as defined by absent or reverse end diastolic flow
   * Biophysical score ≤ 4/10 on 2 occasions
   * Oligohydramnios (deepest vertical pocket less than 2 x 2cm on ultrasound)
   * Other maternal or fetal conditions that would preclude expectant management
2. Known lethal or major fetal anomaly
3. Recent (within 12 months) history of maternal alcoholism or drug dependence
4. Diagnosis of epilepsy
5. Has need for chronic therapy with nonsteroidal anti-inflammatory drugs (NSAIDs) including selective cyclooxygenase (Cox)-2 inhibitors, or unwilling to abstain from use of NSAIDs during the study treatment period (low dose aspirin of 81 mg/day or less allowable)
6. Received within 72 hours or has requirement for heparin; low molecular weight heparins such as enoxaparin or dalteparin; fondaparinux; antiplatelet agents such as clopidogrel, prasugrel, or high dose aspirin (>81 mg/day); Direct Thrombin Inhibitors (DTI) such as dabigatran
7. Pre-existing renal disease, documented pre-pregnancy or in pregnancy prior to 20 weeks gestation (prior to the diagnosis of preeclampsia) or 24 hr urine of ≥0.3 gm/24 hours, documented in pregnancy, prior to 20 weeks gestation or ≥2+ dipstick or ≥ 0.3 Protein Creatinine Ratio (PCR), documented in pregnancy at the last available test prior to 20 weeks gestation. In the case of conflicting results between dipstick, PCR, and timed urine collection tests to work up an episode of proteinuria, the timed urine collection result would supersede other results
8. Multi-fetal pregnancy
9. History of Antiphospholipid antibody syndrome
10. Known hypersensitivity to goat and goat milk proteins
11. Participation in another interventional clinical trial of an investigational, unapproved therapy (drug, biologic, device) within 30 days of consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07-11 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paidas, MD, Principal Investigator — Yale New Haven Hospital
Locations (23):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - University of California at Irvine, Orange, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Oschner Baptist, New Orleans, Louisiana
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Tri-State Maternal Fetal Health, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women & Infants Hospital, Providence, Rhode Island
  - Erlanger Medical Center, Chattanooga, Tennessee
  - University Texas Medical Branch, Galveston, Texas
  - University of Texas Houston School of Medicine, Houston, Texas
  - Intermountain Health, Murray, Utah
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paidas MJ, Tita ATN, Macones GA, Saade GA, Ehrenkranz RA, Triche EW, Streisand JB, Lam GK, Magann EF, Lewis DF, Dombrowski MP, Werner EF, Branch DW, Habli MA, Grotegut CA, Silver RM, Longo SA, Amon E, Cleary KL, How HY, Novotny SR, Grobman WA, Whiteman VE, Wing DA, Scifres CM, Sibai BM. Prospective, randomized, double-blind, placebo-controlled evaluation of the Pharmacokinetics, Safety and Efficacy of Recombinant Antithrombin Versus Placebo in Preterm Preeclampsia. Am J Obstet Gynecol. 2020 Nov;223(5):739.e1-739.e13. doi: 10.1016/j.ajog.2020.08.004. Epub 2020 Aug 8. PMID 32780999
- [Derived] Cotten CM. Adverse consequences of neonatal antibiotic exposure. Curr Opin Pediatr. 2016 Apr;28(2):141-9. doi: 10.1097/MOP.0000000000000338. PMID 26886785

RESULTS

PARTICIPANT FLOW:
Period: Maternal Follow-up (ITT Population)
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9%
Started | 62 | 58
Completed | 59 | 51
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — declined to see site staff | 0 | 1
Not completed — didn't return to site (f/u elsewhere) | 0 | 1
Period: Neonatal Follow-up (Safety Population)
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9%
Started | 60 | 54
Completed | 56 | 50
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 3 | 2
Not completed — delivered at another hospital | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9% | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (6.1) | 29.3 (6.7) | 29.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 56 | 48 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 27 | 54
  White | 29 | 30 | 59
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 62 | 58 | 120
Gestational Age at Randomization [Mean (Standard Deviation); unit: weeks] | 27.18 (1.96) | 27.34 (2.06) | 27.25 (2.00)
Type of Preeclampsia [Count of Participants; unit: Participants]
  Preeclampsia | 39 | 32 | 71
  Superimposed Preeclampsia | 23 | 26 | 49
Parity (number of previous live births) [Count of Participants; unit: Participants]
  0 | 37 | 16 | 53
  1 | 14 | 20 | 34
  2 | 6 | 11 | 17
  3 | 4 | 4 | 8
  4 | 1 | 6 | 7
  5 | 0 | 1 | 1
  >5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Increase in Gestational Age in Days
Description: Increase in gestational age is defined as the gestational age at delivery minus the gestational age at randomization.
Time Frame: Subjects will continue on study drug until maternal and/or fetal indications for delivery necessitate cessation of expectant management or until 34 0/7 weeks of gestation.
Population: ITT
Measure: Median (Full Range); unit: days
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9%
Number analyzed (Participants) | 62 | 58
days | 5.0 [0 to 75] | 6.0 [0 to 85]

2. Secondary Outcome: Composite Measure of Specific Fetal and Neonatal Outcomes Based on Protocol Defined 5-point Scale (Scores of 0 to 4)
Description: Composite score was calculated based on the following fetal and neonatal events: bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH), cystic periventricular leucomalacia (PVL), retinopathy of prematurity (ROP), late Sepsis, necrotizing enterocolitis (NEC) and mortality (fetal and neonatal). The endpoint is measured on a 5 point scale where 0 represents no outcomes experienced and no mortality, and 4 represents death, as shown below. Should the same outcome occur more than once, it will only be counted once.
  Score Outcome 0 No events, no mortality
  1. One event, no mortality
  2. Two events, no mortality
  3. Three or more events, no mortality
  4. Death
Time Frame: Neonatal outcomes were assessed from birth until the later of 36 weeks (wks) Post Menstrual Age (PMA) and the 36 wks PMA visit, or through the 4-6 weeks post-delivery visit (if both 36 wks PMA and the 36 wks PMA visit occurred < 28 days post delivery)
Population: ITT
Measure: Mean (Standard Deviation); unit: scores on a scale of 0 to 4
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9%
Number analyzed (Participants) | 60 | 56
scores on a scale of 0 to 4 | 0.7 (1.0) | 0.6 (0.9)

3. Other Pre Specified Outcome: Number of Participants Experiencing Individual Maternal, Perinatal and Neonatal Outcomes and Number of Participants Who Avoided All Neonatal Morbidity and Mortality
Description: Maternal and fetal/neonatal outcomes of specific interest were defined in the protocol. Maternal subjects were assessed through 4-6 weeks post delivery to determine if outcomes had occurred. Neonatal outcomes were assessed from birth until 36 weeks post menstrual age, or through the 4-6 week post delivery visit (if 36 weeks PMA occurs <28 days following delivery). A second fetal/neonatal composite outcome was the avoidance of fetal/neonatal mortality and neonatal morbidity [BPD, IVH grade ≥ 3, cystic PVL, ROP stage ≥ 3, late sepsis, and NEC (Bell's stage ≥ 2)].
Time Frame: Maternal-till 4-6 weeks post delivery.Neonatal -birth until the later of 36 weeks PMA and the 36 weeks PMA visit, or through the 4-6 weeks post-delivery visit (if both 36 weeks PMA and the 36 weeks PMA visit occurred less than 28 days following delivery).
Population: ITT
Measure: Number; unit: participants
Arm/Group | Recombinant Human Antithrombin (ATryn) | Normal Saline 0.9%
Number analyzed (Participants) | 62 | 58
participants
  Maternal Death | 0 | 0
  Maternal Eclamptic Seizure | 0 | 1
  Maternal Myocardial Infarction | 0 | 0
  Maternal Cerebrovascular Accident | 0 | 0
  Maternal Transient Ischemic Attack | 0 | 0
  Maternal Progressive Renal Insufficiency | 2 | 0
  Maternal Thrombocytopenia (without HELLP) | 8 | 2
  Maternal HELLP | 2 | 0
  Maternal DIC | 0 | 0
  Maternal Pulmonary Edema | 2 | 4
  Maternal Placental Abruption | 0 | 0
  Maternal Severe Intra and Post-Partum Hemorrhage | 2 | 0
  Maternal VTE Including DVT and Pulmonary Embolism | 1 | 2
  Fetal Death (including stillbirth) | 0 | 0
  Neonatal Death | 3 | 2
  Fetal and neonatal death | 3 | 2
  Neonatal Small for Gestational Age (SGA) <10% | 12 | 9
  Neonatal Respiratory Distress Syndrom (RDS) | 59 | 51
  Neonatal Bronchopulmonary Dysplasia (BPD) | 22 | 20
  Neonatal Retinopathy of Prematurity stage >= 3 | 0 | 0
  Neonatal Necrotizing Enterocolitis-Bell's gr >= 2 | 1 | 2
  Neonatal Intraventricular Hemorrhage gr >= 3 | 3 | 1
  Neonatal Cystic Periventricular Leucomalacia | 2 | 1
  Neonatal Early Sepsis | 0 | 0
  Neonatal Late Sepsis | 2 | 4
  Neonatal Meningitis | 0 | 1
  Avoidance of neonatal morbidity and mortality | 36 | 33

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of obtaining informed consent until completion of the study. AEs in the mother, while pregnant and after delivery, including those affecting the fetus, were collected up to and including the last scheduled visit, 4-6 weeks after delivery. Serious AEs (SAEs) in the neonate were collected from day of birth to the last neonate assessment, 36 weeks post-menstrual age or 4-6 week post-delivery (if 36 weeks PMA occurred < 28 days following delivery).
Description: Note: AEs are presented at the subject level and non-serious AE table below also includes serious AEs. Note: Initially, investigators were instructed to report all neonatal outcomes of interest (OOI) as SAEs. This requirement was removed under Protocol Amendment 4 (approximately 60% of the population). Neonatal OOI continued to be captured as outcomes but were only reported as SAEs if they met the criteria for seriousness outlined in the protocol, as determined by the investigator.
Groups:
- Maternal/Fetal Safety Population: ATryn: Subjects treated with Recombinant human antithrombin (ATryn):
  ATryn 250 mg loading dose over 15 minutes, immediately followed by continuous infusion of 2000 mg per 24 hours. Total daily dose is 2250 mg for the first day and 2000 mg on subsequent days
- Maternal/Fetal Safety Population: Placebo (Normal Saline 0.9%): Subjects treated with Placebo; Placebo (Normal Saline 0.9%, matched for volume of active treatment) consisting of a loading dose over 15 minutes followed by continuous infusion.
- Neonatal Safety Population: ATryn: Neonates born to mothers treated with Recombinant Human Antithrombin (ATryn)
- Neonatal Safety Population: Placebo: Neonates born to mothers treated with placebo (Normal Saline 0.9%)
Arm/Group | Maternal/Fetal Safety Population: ATryn | Maternal/Fetal Safety Population: Placebo (Normal Saline 0.9%) | Neonatal Safety Population: ATryn | Neonatal Safety Population: Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/54 | 3/60 | 2/54
Serious Adverse Events (participants affected / at risk) | 10/60 | 11/54 | 32/60 | 24/54
Other Adverse Events (participants affected / at risk) | 60/60 | 53/54 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal/Fetal Safety Population: ATryn (N=60) | Maternal/Fetal Safety Population: Placebo (Normal Saline 0.9%) (N=54) | Neonatal Safety Population: ATryn (N=60) | Neonatal Safety Population: Placebo (N=54)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal Wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Persistent foetal circulation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Neonatal intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Meningitis neonatal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis neonatal (Infections and infestations) | 0 | 0 | 3 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 3 | 1
Periventricular leukomalacia (Nervous system disorders) | 0 | 0 | 2 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 5 | 3
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 9
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 26 | 21
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory tract haemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 0 | 1 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal/Fetal Safety Population: ATryn (N=60) | Maternal/Fetal Safety Population: Placebo (Normal Saline 0.9%) (N=54) | Neonatal Safety Population: ATryn (N=0) | Neonatal Safety Population: Placebo (N=0)
Hypertension (Vascular disorders) | 32 | 25 | 0 | 0
Headache (Nervous system disorders) | 24 | 19 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 20 | 12 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 0 | 0
Infusion site extravasation (General disorders) | 4 | 15 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Oedema peripheral (General disorders) | 4 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 4 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0
Pyrexia (General disorders) | 2 | 4 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0
Vision blurred (Eye disorders) | 1 | 3 | 0 | 0
Platelet count decreased (Investigations) | 1 | 3 | 0 | 0
Postpartum depression (Psychiatric disorders) | 1 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0

LIMITATIONS AND CAVEATS:
Note: 6 subjects (2 in the Recombinant Human Antithrombin (ATryn) group and 4 in the placebo group) were randomized but received no treatment. These subjects are included in the ITT population but not the maternal safety population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site may publish the results of the study after the multi-center publication or 18 months after the sponsor's final evaluation of all study data from all sites, whichever occurs first.

Up to 90 days prior to submitting a manuscript or prior to any public presentation, a copy of the abstract, manuscript, or presentation will be provided to Sponsor by the Site for review and comment. Sponsor shall have said 90 day period to respond to the Site with comments.